CLINICAL TRIAL: NCT01212094
Title: Double Blind Combination of Rituximab by Intravenous and Intrathecal Injection Versus Placebo in Patients With Low-Inflammatory Secondary Progressive Multiple Sclerosis (RIVITaLISe)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The efficacy on CSF biomarkers failed to reach criteria for continuation of the trial
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 100212; 10-N-0212
Expanded Access: Available
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Multiple Sclerosis
Keywords: Rituximab; Multiple Sclerosis; Intrathecal; MS; Secondary-Progressive Multiple Sclerosis; SP-MS
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive | interventions — Rituximab; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rituximab (Experimental): Patients received 25mg of rituximab into the CSF and 200mg of rituximab intravenously at Month 0, followed by additional 200mg of rituximab intravenously at Month 0.5 and another 25mg of rituximab into CSF at months 1.5 and 12.
  Interventions: Drug: Rituximab
- Placebo (Placebo Comparator): Patients received normal saline into the CSF and intravenously at Month 0, followed by additional normal saline intravenously at Month 0.5 and another dose of normal saline into CSF at months 1.5 and 12.
  Interventions: Other: normal saline
- Baseline (No Intervention): Patients in their first year baseline prior to study drug phase

INTERVENTIONS:
Drug: Rituximab
  Arms: Rituximab
Other: normal saline — normal saline
  Other Names: saline
  Arms: Placebo

SUMMARY:
Background:

- Secondary-progressive multiple sclerosis (SP-MS) is the chronic phase of multiple sclerosis (MS). The majority of people who have relapsing-remitting MS eventually develop SP-MS. There are currently no effective treatments for SP-MS. Researchers are interested in determining whether the drug rituximab, which is used to treat rheumatoid arthritis and some types of cancer, is able to target certain white blood cells that are thought to play a role in the progression of SP-MS. To ensure that the rituximab will reach the brain and spinal cord, participants will receive it by intravenous drip and by intrathecal injection (through a lumbar puncture into the cerebrospinal fluid).

Objectives:

- To evaluate the safety and effectiveness of combined intravenous and intrathecal rituximab in individuals with secondary-progressive multiple sclerosis.

Eligibility:

- Individuals between 18 and 65 years of age who have been diagnosed with SP-MS and have been off any form of immunosuppressive therapy for at least 3 months.

Design:

- The study will involve a 1-year pretreatment baseline series of visits, followed by a 2-year treatment period. Participants will provide blood samples throughout treatment as directed by the study researchers, and additional studies may be performed during the study period if participants consent to further investigation.

DETAILED DESCRIPTION:
Objective: The primary goal of this study is to define the safety and efficacy of combined systemic and intrathecal (IT) B cell-depleting therapy (i.e. anti-CD20, rituximab) in patients with secondary-progressive multiple sclerosis (SP-MS). The secondary goals of this study are to collect longitudinal data to help identify the most sensitive outcome measures and trial design for future Phase II trials for SP-MS patients and to investigate the mechanism of action of rituximab on the human immune system.

Study Population: Patients with SP-MS and mild to moderate level of clinical disability, who have no medical contraindication to IT or intravenous (IV) administration of rituximab.

Design: This is double blind, placebo-controlled, single center, baseline versus treatment, Phase I/II clinical trial of IV and IT rituximab in SP-MS patients.

Outcome Measures: Quantitative neuroimaging measures of central nervous system (CNS: i.e. brain and spinal cord) tissue destruction and clinical and functional (i.e. electrophysiological) measures of neurological disability will be collected every 6-12 months. Additionally, biomarkers focusing on analysis of cerebral spinal fluid (CSF) B cells and immunological responses to EBV will be collected at baseline and during treatment. The trial is currently powered using progression of brain atrophy as detected by SIENA methodology as the primary outcome measure. However, this may not be the most sensitive outcome available. In recognition of this, the trial has an adaptive design: it incorporates analysis of the progression of CNS tissue destruction, as measured by quantitative MRI markers, and clinical/paraclinical markers, defined as secondary outcome measures, in the first 30 enrolled patients during the year long pre-treatment baseline prior to randomization. All defined outcome measures collected in the first 30 enrolled patients will be transformed into z-scores and compared for the robustness of longitudinal change over the coefficient of variation. As a result, the primary outcome measure of this trial will be the comparison of individualized rates of brain atrophy progression between the rituximab and placebo groups after 2 years of treatment; unless the predetermined analysis establishes that one of the secondary outcome measures has a higher z-score than the brain atrophy measurement. In this case, the primary outcome would be the efficacy of rituximab versus placebo in inhibiting patient-specific slopes of functional or structural deterioration as measured by this more sensitive biomarker of CNS tissue destruction.

Trial also included interim analysis for the efficacy of B cell depletion from the intrathecal compartment with pre-defined stopping criteria for futility: if less than 50% of intrathecal B cells were depleted by active treatment (measured by <25% decrease in CSF CXCL13 and <50% increase in CSF BAFF), then trial was deemed to be underpowered to demonstrate efficacy on clinical or MRI outcomes and would be stopped.

ELIGIBILITY:
* INCLUSION CRITERIA:

MS as defined by the modified McDonald s criteria (Polman, Reingold et al. 2005)

SP-MS as documented by lack of MS relapse for the past 1 year and non-remitting/sustained (> 3 months) progression of disability

Age 18-65, inclusive, at the time of the first screening baseline visit

EDSS 3.0 to 7.0, inclusive, at the time of the first screening baseline visit

Able to provide informed consent

Willing to participate in all aspects of trial design and follow-up

Lack of CEL on all MRIs performed within the last 12 months or if patient has CEL, then documentation that they tried and failed or could not tolerate FDA approved disease modifying therapies (DMTh)

Not receiving any DMTh (such as IFN-beta preparation, glatiramer acetate, corticosteroid, natalizumab, fingolimod, immunosuppressive agents or experimental therapeutics) for a period of at least 1 month before enrollment in the study, allowing for at least a 1-year

period off therapy prior to the first study dose

Agreeing to commit to the use of a reliable/accepted method of birth control (i.e. hormonal contraception (birth control pills, injected hormones, vaginal ring), intrauterine device, barrier methods with spermicide (diaphragm with spermicide, condom with spermicide) or they have undergone surgical sterilization (such as hysterectomy, tubal ligation, or vasectomy)) during enrollment in the study and through 12 months after the last dose of study drug

EXCLUSION CRITERIA:

RR-MS or PP-MS

Evidence of clearly documented MS relapse within the last 1 year

Alternative diagnoses that can explain neurological disability and MRI findings

Clinically significant medical disorders that, in the judgment of the investigators could cause CNS tissue damage, limit its repair, expose the patient to undue risk of harm or prevent the patient from completing the study (such as, but not limited to cerebrovascular disease, ischemic cardiomyopathy, clotting disorder, brittle diabetes, neurodegenerative disorder)

Pregnant or breastfeeding female

History or sign of congenital or acquired immunodeficiency or chronic infections, such as HIV/AIDS, Hepatitis A, B or C, HTLV-1 carrier and others that would expose patient to risks of pathogen reactivation associated with rituximab treatment

Abnormal screening/baseline blood tests exceeding any of the limits defined below:

1. Serum alanine transaminase or aspartate transaminase levels which are greater than three times the upper limit of normal values.
2. Total white blood cell count < 3 000/mm(3)
3. Platelet count < 85 000/mm(3)
4. Serum creatinine level > 2.0 mg/dl and eGFR (glomerular filtration rate) < 60
5. Serological evidence of HIV, HTLV-1 or active hepatitis A, B or C
6. Positive pregnancy test
7. Positive CSF or serum quantitative PCR for JC virus on CSF collected from the baseline spinal tap (test will be performed by CLIA certified laboratory of Gene Major, NINDS)
8. Total serum IgG < 600mg/dl (nl 642-1730mg/dl) or total serum IgM < 30mg/dl (nl 34-342mg/dl) as these Ig deficiencies would suggest underlying abnormalities with B cell function/maturation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bibiana Bielekova, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kosa P, Komori M, Waters R, Wu T, Cortese I, Ohayon J, Fenton K, Cherup J, Gedeon T, Bielekova B. Novel composite MRI scale correlates highly with disability in multiple sclerosis patients. Mult Scler Relat Disord. 2015 Nov;4(6):526-35. doi: 10.1016/j.msard.2015.08.009. Epub 2015 Aug 28. PMID 26590659
- [Derived] Kosa P, Ghazali D, Tanigawa M, Barbour C, Cortese I, Kelley W, Snyder B, Ohayon J, Fenton K, Lehky T, Wu T, Greenwood M, Nair G, Bielekova B. Development of a Sensitive Outcome for Economical Drug Screening for Progressive Multiple Sclerosis Treatment. Front Neurol. 2016 Aug 15;7:131. doi: 10.3389/fneur.2016.00131. eCollection 2016. PMID 27574516
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-N-0212.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject received an open label study drug under a compassionate use amendment of the protocol. This subject is not reflected in the data analysis for the primary or secondary outcome measures.
Groups:
- Placebo: Group administered placebo
- Rituximab: Group administered active drug
Period: Year 1: Baseline Monitoring
Arm/Group | Baseline | Placebo | Rituximab
Started | 43 | 0 | 0
Completed | 27 | 0 | 0
Not Completed | 16 | 0 | 0
Not completed — Study terminated | 7 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 0 | 0
Not completed — Started on DMT | 2 | 0 | 0
Period: Years 2 & 3: Treatment Randomization
Arm/Group | Baseline | Placebo | Rituximab
Started | 0 | 9 | 18
Completed | 0 | 5 | 7
Not Completed | 0 | 4 | 11
Not completed — Study terminated | 0 | 4 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Baseline: Patients in their first year baseline prior to treatment phase
- Total: Total of all reporting groups
Arm/Group | Placebo | Rituximab | Baseline | Total
Number analyzed (Participants) | 9 | 18 | 16 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 18 | 16 | 43
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 11 | 22
  Male | 7 | 9 | 5 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 1 | 4
  White | 6 | 18 | 13 | 37
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Secondary Outcome: Analysis of Changes in CSF B Cell Numbers Between Rituximab and Placebo
Description: This outcome is for interim analysis of the efficacy of B cell depletion from the CSF 3 months after giving rituximab or placebo into the cerebrospinal fluid (CSF). It compares absolute numbers of CSF B cells calculated as proportion of B cells (identified from flow cytometry data) in all immune cells measured in 50-fold concentrated CSF. We averaged two time-points before treatment (CSF collected 1 year apart, at month -12 and month 0) and compared it to the single time-point (month 3), which was 3 months from the initiation of drug dosing.
Time Frame: 3 months
Population: These patients were analyzed for the interim analysis for the efficacy of B cell depletion. Trial stipulated stopping criteria for futility.
Measure: Median (Inter-Quartile Range); unit: percentage of b cell depletion
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 9 | 14
percentage of b cell depletion | -21.6 [-70.4 to 25.4] | -50.7 [-83.3 to 49.3]

2. Primary Outcome: Analysis of Changes in CSF CXCL13 Induced by Active Treatment (Rituximab) Measured 3 Months After 1st Drug Administration
Description: This outcome is for interim analysis of the efficacy of B cell depletion from the CSF 3 months after giving rituximab or placebo into the cerebrospinal fluid (CSF). It compares concentration of chemokine CXCL13 before and 3 months after administration of drug into the CSF. We averaged two time-points before treatment (CSF collected 1 year apart, at month -12 and month 0) and compared it to the single time-point (month 3), which was 3 months from the initiation of drug dosing. CXCL13 is released by activated B cells, T cells and by follicular dendritic cells and has been linked previously with MS inflammation in the brain and spinal cord. The protocol-stipulated threshold for trial continuation was at least 25% decrease in CSF CXCL13 induced by active treatment with significance level p=0.025.
Time Frame: 3 months
Population: For the decision to continue trial, only change from baseline to 3 months post-treatment was analyzed in patients who received active drug
Measure: Median (Inter-Quartile Range); unit: percentage of b cell depletion
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 9 | 14
percentage of b cell depletion | 0 [0 to 0] | -11.9 [-100 to 0]

3. Primary Outcome: Analysis of Changes in CSF BAFF Induced by Active Treatment (Rituximab) Measured 3 Months After 1st Drug Administration
Description: This outcome is for interim analysis of the efficacy of B cell depletion from the CSF 3 months after giving rituximab or placebo into the cerebrospinal fluid (CSF). It compares concentration of B-cell activating factor (BAFF) before and 3 months after administration of drug into the CSF. We averaged two time-points before treatment (CSF collected 1 year apart, at month -12 and month 0) and compared it to the single time-point (month 3), which was 3 months from the initiation of drug dosing. BAFF is consumed by B cells, therefore effective B cell depletion increases levels of BAFF. The protocol-stipulated threshold for trial continuation was at least 50% increase in CSF BAFF induced by active treatment with significance level p=0.025.
Time Frame: 3 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage of BAFF change
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 9 | 14
percentage of BAFF change | 4 [-11.2 to 20.5] | 20.9 [-0.3 to 24.9]

4. Secondary Outcome: Expanded Disability Status Scale (EDSS)
Description: Trial was closed prematurely and therefore formal statistical analysis of the acquired clinical outcomes was not performed. EDSS is a clinical rating scale for disability ranging from 0 (normal neurological exam) to 10 (death due to MS) in half point increments.
Time Frame: 24 months
Population: Only 5 patients per group finished Month 24 following 2 years in study drug phase of trial (2 IV doses and 3 IT doses) at the time the study was terminated for futility
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 5 | 5
units on a scale | 6.5 [6.5 to 7] | 6.5 [6.5 to 6.5]

5. Secondary Outcome: Scripps Neurological Rating Scale (NRS)
Description: NRS is a quantitative assessment based on 22 parameters of the neurological exam with scores ranging from maximum of 100 (normal neurological exam) to a minimum of -10 (death due to MS). The higher the score, the better the patient's level of function.
  trial was closed prematurely and therefore formal statistical analysis of the acquired clinical outcomes makes no sense
Time Frame: 24 months
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 5 | 5
units on a scale | 53 [52 to 55] | 53 [53 to 61]

6. Secondary Outcome: Timed 25 Foot Walk
Description: Measure of mobility and leg function based on a timed 25 foot walk. Patient is directed to walk as quickly as possible, with or without an assitive device, to one end of a 25foot course and this is repeated for a total of 2 times. The score is the average of the two completed trials.
  Trial was closed prematurely and therefore formal statistical analysis of the acquired clinical outcomes makes no sense
Time Frame: 24 months
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 5 | 5
seconds | 18.7 [11.7 to 32.7] | 19.1 [8.7 to 27.2]

7. Secondary Outcome: 9-Hole Peg Test
Description: Measure of upper extremity (arm and hand) function where patients are asked to pick up one peg at a time, using one hand only, and putting them into the holes as quickly as possible until all the holes are filled and then removing them one at a time as quickly as possible. The dominant and non-dominant hands are tested twice. The time limit per trial is 5 minutes.
  Trial was closed prematurely and therefore formal statistical analysis of the acquired clinical outcomes makes no sense
Time Frame: 24 months
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 5 | 5
seconds | 25.1 [23.4 to 48.8] | 36.7 [36.1 to 45.9]

8. Secondary Outcome: Multiple Sclerosis Functional Composite (MSFC)
Description: The MSFC is a three-part standardized assessment tool that measures arm, leg, and cognitive function. The scoring is based on the average Z-score for all three parts of the the assessment.
Time Frame: 24 months
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Z score
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 5 | 5
Z score | -0.7 [-1.2 to 0.2] | -0.9 [-2.3 to -0.7]

9. Secondary Outcome: EDSS
Description: as for outcome 4
Time Frame: 0 months
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 5 | 5
units on a scale | 6.5 [6.5 to 6.5] | 6.5 [6.0 to 6.5]

10. Secondary Outcome: Scripps Neurological Rating Scale (NRS)
Description: as for outcome 5
Time Frame: 0 Months
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 5 | 5
units on a scale | 57 [54 to 60] | 59 [52.3 to 62.5]

11. Secondary Outcome: Timed 25 Foot Walk
Description: as for outcome 6
Time Frame: 0 months
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 5 | 5
seconds | 11.9 [8.2 to 29.8] | 11.7 [7.6 to 23.6]

12. Secondary Outcome: 9-Hole Peg Test
Description: as for outcome 7
Time Frame: 0 months
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 5 | 5
seconds | 33.7 [25.8 to 44.5] | 38.3 [28.8 to 42.4]

13. Secondary Outcome: Multiple Sclerosis Functional Composite (MSFC)
Description: as for outcome 8
Time Frame: 0 Months
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Z score
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 5 | 5
Z score | -0.8 [-1.1 to -0.5] | -0.9 [-1.6 to -0.4]

ADVERSE EVENTS:
Time Frame: 36 months
Description: First 12 months (Month -12 to Month 0), all patients were untreated; next 24 months (Month 0 to Month 24) patients were randomized to placebo or active treatment
Groups:
- Placebo: Placebo group
- Rituximab: Group who got active drug
Arm/Group | Placebo | Rituximab | Baseline
Serious Adverse Events (participants affected / at risk) | 4/9 | 4/18 | 0/43
Other Adverse Events (participants affected / at risk) | 9/9 | 18/18 | 8/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | Rituximab (N=18) | Baseline (N=43)
Elevated Blood Sugar (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Post LP Headache (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Neck and Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cognitive Decline (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Gallstones (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | Rituximab (N=18) | Baseline (N=43)
Tachycardia (Cardiac disorders) | 2 (2) | 4 (4) | 0 (0)
anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Nausea/Vomitting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
UTI (Renal and urinary disorders) | 5 (8) | 5 (11) | 0 (0)
kidney stone (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0)
Enhancing brain lesion (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 7 (8) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 5 (7) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Elevated Liver Enzymes (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Teeth Cracking (General disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lipoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Trigeminal Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
fever (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
bunionectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Fungal Infection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Shoulder Dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
laceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Torn Meniscus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dislocated Shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Medication Refill (General disorders) | 0 (0) | 0 (0) | 1 (1) — event was classified as an SAE by the IRB however no hospitalization was needed and the event did not result in other serious outcomes.

LIMITATIONS AND CAVEATS:
The trial was closed prematurely for futility, because pre-determined interim analysis demonstrated that selected dosing led to <50% depletion of B cells from the brain/spinal cord. Therefore, only 5 patients per group finished trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No